CLINICAL TRIAL: NCT01390935
Title: SUrvey of Guideline Adherence for Treatment of Systolic Heart Failure in Real WorldMulticenter, Retrospective Observation Study in Korea
Brief Title: SUrvey of Guideline Adherence for Treatment of Systolic Heart Failure in Real World
Acronym: SUGAR
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114993
Record Dates: First submitted 2011-06-09; First posted 2011-07-11 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Heart Failure, Congestive
Keywords: guideline adherence; systolic heart failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — Guideline Adherence; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- systolic heart failure: EF under 45%
  Interventions: Other: guideline adherence

INTERVENTIONS:
Other: guideline adherence — guideline adherence of physician
  Other Names: ACEI; ARB; BB; aldosterone antagonist

SUMMARY:
The purpose of this study is to survey the guideline compliance of the cardiologists in the treatment of systolic heart failure in Korea

DETAILED DESCRIPTION:
Major improvement in the medical management of CHF has been achieved in the past decades.

But there is no doubt that prognosis of heart failure patients remains poor. The compliance to the standard treatment can be one of reasons. But very little data concerning this in Korea is available.

ELIGIBILITY:
Inclusion Criteria:

* Subjects admitted to hospital with systolic heart failure(LVEF under 45%) in 2009
* Subjects, age 20 or/and above
* Subjects admitted to hospital (emergency area, to internal medicine or to cardiology wards, CCU or intensive care) with dyspnea and verification of heart failure based on following criteria;
* Symptoms typical of heart failure : breathlessness at rest or on exercise, fatigue, tiredness, ankle swelling and Signs typical of heart failure : tachycardia, tachypnoea, pulmonary rales, pleural effusion, raised jugular venous pressure, peripheral oedema, hepatomegaly
* Objective evidence of a structural or functional abnormality of the heart at rest : cardiomegaly, third heard sound, cardiac murmurs, abnormality on the echocardiogram, raised natriuretic peptide concentration

Exclusion Criteria:

* Subject who expired during hospitalization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: admission for systolic heart failure in general hospital
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Mean of modified Guideline Adherence Indicator(mGAI-3) | 1year
  Modified percentage based on each participant's condition

SECONDARY OUTCOMES:
Percentage of participants with each class drug prescribed | 1year
  ARB, BB, ACE-I, aldosterone antagonist
Percentage of participants with daily target dose reached | 1year
  ARB, BB, ACE-I, aldosterone antagonist
Percentage of all cause mortality | 1year
  All cause mortality in 1-year after treatment of systolic heart failure
Percentage of All cause hospitalization | 1year
  All cause hospitalization in 1-year after treatment of systolic heart failure
Mean of mortality or rehospitalization rate according to mGAI-3 | 1year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea